CLINICAL TRIAL: NCT05931302
Title: Initial Staging of Lobular Breast Carcinoma: Head to Head Comparison of 68Ga-FAPI-46 and 18F-FDG PET/CT
Acronym: GALILEE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Institut Curie (Other); Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-CHITS-006
Record Dates: First submitted 2023-06-16; First posted 2023-07-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Lobular Breast Carcinoma
Keywords: 68Ga-FAPI-46; 18F-FDG PET; FAPα; staging
MeSH Terms: conditions — Carcinoma, Lobular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI-46 PET scan + 18-FDG PET scan (Experimental)
  Interventions: Diagnostic Test: 68Ga-FAPI-46 PET scan

INTERVENTIONS:
Diagnostic Test: 68Ga-FAPI-46 PET scan — 68Ga-FAPI-46 is a radiotracer for the detection of Fibroblast Activation Protein (FAP) in cancer patients.
  68Ga-FAPI-46 will be administered intravenously at a dose of 2MBq/kg. Patients will be scanned 60 minutes after administration of 68Ga-FAPI-46.

SUMMARY:
Lobular Breast cancer staging with 18F-fluorodeoxyglucose positron emission tomography (18F-FDG PET) is not optimal due to the poor accumulation of 18F-FDG in the tumour. Through better sensitivity (and specificity), 68Ga-FAPI-46-46 PET should provide a more accurate staging of lobular breast cancer than 18F-FDG PET.

DETAILED DESCRIPTION:
Research hypothesis : Through better sensitivity (and specificity), 68Ga-FAPI-46-46 PET should provide a more accurate staging of lobular breast cancer than 18F-FDG PET. Participants with lobular breast carcinoma will then undergo 18F-FDG and 68Ga-FAPI-46 PET scan.

Primary objective of the study is to compare the sensitivity of 68Ga-FAPI-46 with the sensitivity of 18F-FDG in the detection of lobular breast carcinoma lesions, measured by positron emission tomography (PET). These results will be compared with the histological data collected before or during surgery (conventional histological data and immunohistochemical labeling of FAPα on the sample obtained), clinical follow-up and any results of additional examinations carried out within the usual clinical follow-up of the patients.

Comparison of primary tumor and metastases uptake of 68Ga-FAPI-46 with the uptake of 18F-FDG, radiomic study of 68Ga-FAPI-46 PET and comparative radiomic study of 68Ga-FAPI-46 PET and 18F-FDG PET and comparison of the specificity of 68Ga-FAPI-46 with the specificity of 18F-FDG after a 12-month follow-up will also be performed as secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* ECOG from 0 to 2
* Histological diagnosis of Lobular Carcinoma of the breast based on a breast biopsy
* Patient naïve to any treatment for lobular breast carcinoma
* Women of childbearing age should have an adequate method of contraception
* Patient having voluntarily accepted to participate in the study and signed the informed consent
* Minimum tumor stage IIA
* Sufficient histological material in the biopsy or the surgical specimen, if the biopsy is insufficient

Exclusion Criteria:

* PET scan contraindications: severe claustrophobia, unbalanced diabetes during 18F-FDG PET scans (fasting capillary blood sugar ≥ 11 mmol)
* Hormone therapy started
* 18F-FDG PET scan > 21 days
* Pregnant women, parturients and nursing mothers
* Persons deprived of liberty by a judicial or administrative decision
* Persons admitted to a health or social establishment for purposes other than research
* Adults who are the subject of a legal protection measure or who are unable to express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Number of positive tumor lesions, i.e. confirmed by additional imaging, histopathology/biopsy or response to treatment (on imaging or clinical assessment) | Up to 12 months
  Number of positive tumor lesions of 68Ga-FAPI-46 PET scan in comparison with 18F-FDG PET scan

SECONDARY OUTCOMES:
SUVmaxFAPI and SUVmaxFDG for each target (Standardized Uptake Value) | Up to 21 days
  Comparison of 68Ga-FAPI-46 and 18F-FDG Standardized Uptake Value in the primary tumor and possible metastases
SUVmaxFAPI/reference and SUVmaxFDG/reference activity ratios | Up to 21 days
  Comparison of (SUVmaxFAPI/reference) and (SUVmaxFDG/reference) activity ratios. For the primary tumour, the reference activity will be measured in either the periphery of the lesion or on a homologous healthy tissue. For a vertebral metastasis, the reference activity will be measured in an adjacent healthy vertebra.
MTVFAPI and MTVFDG (Metabolic Tumor Volume) | Up to 21 days
  Comparison of MTVFAPI and MTVFDG in the primary tumor and possible metastases
Number of discrepancies between FAPI and FDG PET scans | Up to 21 days
  Discrepancies (discordant pairs) between 68Ga-FAPI-46 PET scan and 18F-FDG PET scan will be analyzed
Correlation between PET scan and FAPα labeling | Up to 12 months
  Correlation between PET scan results and measurement of the FAPα labeling density on the biopsy
Correlation between PET scan and breast histology | Up to 12 months
  Correlation between PET scans results and standard measurements in breast histology: OR (estrogen receptors), PR (progesterone receptors), HER2 (Human Epidermal Growth Factor Receptor-2), Ki-67 antigen, Ecadherin
Specificity comparison | 12 months
  Specificity of 68Ga-FAPI-46 PET scan will be compared to 18F-FDG PET scan specificity
Correlation between tumor lesion radiomics and histological characteristics | 12 months
  1st order characteristics reflecting the distribution of gray levels determined by radiomics study of 68Ga-FAPI PET scan and 18F-FDG PET scan

CONTACTS AND LOCATIONS:
Overall Officials: Florent Hugonnet, MD, Study Director — Centre Hospitalier Princesse Grace
Locations (1):
- Centre Hospitalier Princesse Grace, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No